CLINICAL TRIAL: NCT05753176
Title: Online 1-Day CBT-Based Workshops for Preventing Postpartum Depression: A Randomized Controlled Trial
Brief Title: Online 1-Day CBT-Based Workshops for Preventing Postpartum Depression
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: RCT1-day CBT to prevent PPD
Record Dates: First submitted 2023-01-26; First posted 2023-03-03 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Postpartum Depression; Postpartum Anxiety
Keywords: cognitive behavioral therapy; CBT; postpartum depression; PPD; randomized controlled trial; RCT
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Intervention Model Description: A parallel-group Ontario-wide RCT with experimental (workshop) and TAU (control) groups will address our objectives. Participants will be randomly assigned in a 1:1 ratio to the treatment or control group.
Who Masked: Outcomes Assessor
Masking Description: Participants and the research coordinator cannot be blinded to group condition though the research assistants sending out 1, 2, and 3 month postpartum follow questionnaires and data analysts will not be aware of group status.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online 1-Day CBT-Based Workshop (Experimental): Participants assigned to the treatment arm will attend a day long CBT-based workshop delivered online by two trained facilitators in addition to receiving usual care.
  Interventions: Behavioral: Online 1-Day Cognitive Behavioural Therapy-Based Workshop
- Treatment as Usual (No Intervention): Participants assigned to the control arm will continue to receive standard prenatal care from their healthcare providers.

INTERVENTIONS:
Behavioral: Online 1-Day Cognitive Behavioural Therapy-Based Workshop — The Online Workshop is a day-long intervention delivered by two trained facilitators (i.e., psychotherapists, social workers, nurses, and/or a psychiatrist) consisting of 6 hours of instruction delivered in 4 modules. The 1st contains information on PPD etiology with a focus on modifiable cognitive risk factors (e.g., negative thoughts, maladaptive core beliefs). The 2nd module focuses on cognitive skills including cognitive restructuring. The 3rd builds behavioural skills such as problem solving, behavioural activation, assertiveness, sleep strategies, and using supports. The final module provides an opportunity for goal setting/action planning. Teaching methods include didactic sections, group exercises, and role-plays. Regular breaks are incorporated. Each participant is given a professionally designed manual to facilitate learning. Participants are also given a list of region-specific PPD resources and a copy of the Canadian Practice Guidelines for the treatment of PPD.
  Arms: Online 1-Day CBT-Based Workshop

SUMMARY:
To conduct a randomized controlled trial (N=408) examining the impact of an online cognitive behavioural therapy (CBT)-based workshop on rates of postpartum depression (i.e., EPDS scores at 2-months postpartum) when added to treatment as usual (TAU) compared to TAU alone.

DETAILED DESCRIPTION:
Postpartum depression affects up to 1 in 5 mothers, however just 15% receive evidence-based treatment. It is associated with negative consequences for women and their families with enormous costs to the healthcare system. Postpartum depression is an ideal candidate for prevention because it is common, the window of opportunity to intervene is clear (pregnancy), and its risk factors are well-established and easily identifiable. Furthermore, women are in frequent contact with the healthcare system during pregnancy and are more motivated to improve their health during this time than at any other time in their lives. Given the high rate of PPD and its adverse effects on mothers and their families, and the relative lack of efficient, effective psychotherapeutic interventions for preventing PPD, safe, novel, and efficient preventive interventions are needed. Since large 1-day workshops appear to successfully treat depression, given the widespread interest and investment of public health units across Canada in maternal and child health, Online 1-Day CBT-Based Workshops for Preventing PPD should be developed and tested for their ability to prevent PPD in Canadian women.

Based on longstanding clinical work with women at high risk for PPD, the development of a successful 1-Day CBT-Based Treatment Workshop for PPD and its delivery in-person and online, and an extensive review of the PPD prevention literature, the investigators developed the content for our prevention workshop as well as an accompanying script and intervention manual for participants in a previous pilot study. This pilot study also assessed feasibility by recruiting 32 women who took part in an online CBT-based workshop and provided feedback on its content, delivery and assessment procedures. The workshop, manual, and study protocol were subsequently refined and our experience recruiting participants in community settings into CBT treatment studies for PPD will be utilized in the current randomized controlled trial (N=408), which is aimed as assessing the effectiveness of these workshops at reducing the likelihood of developing PPD in women at risk.

Objectives of the proposed randomized controlled trial are as follows:

Primary: To determine if Online 1-Day CBT-Based Workshops delivered to pregnant persons with a past history of major depressive disorder (MDD) and added to TAU reduces EPDS scores at 2-months postpartum more than TAU alone and to determine if these workshops reduce the risk of developing PPD (EPDS score ≥13 at 2 months postpartum).

Secondary: To determine if 1-Day CBT-based workshops lead to differences in the common comorbidities of PPD (maternal anxiety, problems with the mother-infant relationship, infant temperament, maternal social support, and maternal perceived stress) between the experimental and control groups.

Tertiary: To determine if 1-Day CBT-based workshops alter trajectories of PPD and its comorbidities from birth to three months postpartum and whether they are cost- effective.

Additional Analyses: A subgroup analysis will be conducted in those participants deemed as being of low socioeconomic status. The investigators will also conduct subgroup analyses to determine whether there are any differences in the magnitude of the treatment effect in participants that are single marital status, have a past history of abuse or have poor social support. Additional subgroup analyses will be conducted in those participants who are first time mothers, those who have generalized anxiety disorder, and those receiving treatment for past depression at baseline.

A prospective randomized controlled trial design will be used to address these objectives. The study will be advertised through our public health and community partners (i.e., midwifery associations) in Ontario, as well as on Facebook and Instagram. Participants will be allocated in a 1:1 ratio to experimental (1-Day CBT Workshop in addition to TAU) or control (TAU alone) groups. Both experimental and control groups will complete data collection at baseline (before completing the 1-Day CBT workshop for experimental group participants), and at 1, 2 and 3 months postpartum.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Currently residing in Ontario, Canada
* Currently in 3rd trimester of pregnancy (28-36 weeks gestation)
* EPDS score >6
* Past history of major depressive disorder (determined using the Mini International Neuropsychiatric Interview (MINI)

Exclusion Criteria:

* positive score on the MINI for a current major depressive episode
* positive score on the MINI subsections of bipolar, psychotic, or borderline personality disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 412 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
EPDS score as a continuous outcome (Total EPDS) and an EPDS score of 13 or more at 2-months postpartum (T3) will serve as co-primary outcomes. | Baseline (T1), 1-month postpartum (T2), 2-months postpartum (T3), and 3-months postpartum (T4)
  Edinburgh Postnatal Depression Scale (EPDS): the gold standard measure of PPD symptoms in clinical practice and research. The EPDS is a self-report 10-item scale scored out of 30 points that measures the severity of depressive symptoms in the past 7 days. Scores are between 0 and 30, with higher scores indicating the presence of more depressive symptoms. Scores of 13 and above indicate depressive illness, or a high risk of developing a depressive disorder. A reduction of four points in the EPDS is recognized as a clinically significant improvement.

SECONDARY OUTCOMES:
Maternal Anxiety (Generalized Anxiety Disorder 7-Item Scale (GAD-7)) | Baseline (T1), 1-month postpartum (T2), 2-months postpartum (T3), and 3-months postpartum (T4)
  The Generalized Anxiety Disorder 7-Item Scale (GAD-7) is a validated 7-item self-report scale that identifies probable cases of generalized anxiety disorder (GAD) and severity of anxiety symptoms, the most common PPD comorbidity that is known to be responsive to CBT. Respondents rate how often they have been bothered by various symptoms by providing a score on a 4-point Likert scale ranging from 'not at all' to 'nearly every day'. A higher score on this scale indicates greater severity of anxiety.
Maternal Social Support (MSPSS) | Baseline (T1), 1-month postpartum (T2), 2-months postpartum (T3), and 3-months postpartum (T4)
  The Multidimensional Scale of Perceived Social Support (MSPSS)MSPSS is a 12-item measure of perceived adequacy of social support from three sources: friends, family and significant other. It is scored using a 5-point Likert scale (0=strongly disagree, 5=strongly agree). Higher scores indicated higher perceived adequacy of social support.
Maternal Perceived Stress (Perceived Stress Scale (PSS)) | Baseline (T1), 1-month postpartum (T2), 2-months postpartum (T3), and 3-months postpartum (T4)
  The Perceived Stress Scale (PSS) is one of the most widely used psychological instruments for measuring the perception of stress. The PSS measures the degree to which situations are appraised as stressful and items tap how unpredictable, uncontrollable, and overloaded respondents find their lives. The questions in this scale ask about feelings and thoughts experienced during the last month, and respondents are asked to indicate how often they felt or thought a certain way on a 5-point Likert scale ranging from 0=never to 4=very often. Scores range from 0 to 40 with scores between 0-13 considered low stress, 14-26 considered moderate stress, and 27-40 considered high perceived stress.
Problems with the Mother-Infant Relationship (Postpartum Bonding Questionnaire (PBQ)) | 1-month postpartum (T2), 2-months postpartum (T3), and 3-months postpartum (T4)
  The Postpartum Bonding Questionnaire (PBQ) is a 25-item maternal-report measure that assesses four aspects of maternal-infant relations: (1) bonding, (2) rejection and anger towards the infant, (3) infant-focused anxiety and (4) incipient abuse. Subscales 1-3 will be explored as a continuous outcome using subscale total score. Each item is scored on a scale of 0-5, with higher scores suggestive of more problems. Mother-infant bonding will be measured as a continuous and dichotomous outcome, using cut-off scores for each subscale indicating bonding disorders. Cutoff values of 12 for the bonding subscale, 17 for rejection and anger, and 10 for infant-focused anxiety have been proposed to define bonding disorders in each category.
Infant Temperament (Infant Behaviour Questionnaire-Revised (IBQ-R)) | 3-months postpartum (T4)
  The IBQ-R is a 91-item self-report, gold-standard measure of infant temperament. This measure is completed by mothers who report on their infant's behaviour and temperament. How often a mother observes each behaviour in a week is measured on 7-point scale from 1 (never) to 7 (always). This scale assesses temperament on 14 subscales: Activity Level, Distress to Limitations, Approach, Fear, Duration of Orienting, Smiling and Laughter, Vocal Reactivity, Sadness, Perceptual Sensitivity, High Intensity Pleasure, Low Intensity Pleasure, Cuddliness, Soothability, and Falling Reactivity/Rate of Recovery from Distress. Respondents indicate how often the infant did each behaviour during the past seven days by choosing a number between 1 (never) to 7 (always).

OTHER OUTCOMES:
Cost-Effectiveness - Healthcare Costs | Baseline (T1) (mother only) and 3-months postpartum (T4) (infant and mother)
  Healthcare resource utilization data (including mental health service use) will be collected using a questionnaire based on the Canadian Community Health Survey and the Service Use and Resources Form, adapted for the postpartum period and used in previous PPD research. Resources consumed over the trial period from the perspective of the public health care payer will be measured. Corresponding unit costs will be calculated using provincial or other standard billing rates. Participants will provide information on resource use including diagnoses, procedures, medications, hospital stays, physician and ER visits, and use of other healthcare providers. Separate data will be collected for healthcare resources used by the mother and healthcare resources used by the infant.
Cost Effectiveness - Quality-Adjusted Life Year | Baseline (T1), 1-month postpartum (T2), 2-months postpartum (T3), and 3-months postpartum (T4)
  Cost-effectiveness will be measured using incremental cost per quality-adjusted life year ratio.
  Quality-Adjusted Life Year (QALY): The EQ-5D-5L is a utility-based health-related quality of life instrument consisting of five questions covering depression/anxiety, usual activities, self-care, pain/ discomfort, and mobility. Its Canadian scoring algorithm will be used to convert the five responses to health utility at baseline, and one, two, and three months postpartum. For each participant, a QALY will be calculated by multiplying the health utility for the matching time period (i.e., the area under the curve approach).
Client Satisfaction (Client Satisfaction Questionnaire (CSQ-8)) | 1 week post-intervention in the experimental arm
  Intervention participants only. An 8-item scale that measures and assesses consumer satisfaction with health and human services. Items are scored on a 4-point scale and total scores range from 8-32, with higher scores indicating greater satisfaction.
Client Satisfaction (Client Satisfaction Questionnaire (CSQ-8)) | 3-months postpartum (T4)
  Intervention participants only. An 8-item scale that measures and assesses consumer satisfaction with health and human services. Items are scored on a 4-point scale and total scores range from 8-32, with higher scores indicating greater satisfaction.
Cognitive Behavioural Therapy Skills Acquisition | 1-month postpartum (T2) and 3-months postpartum (T4)
  Cognitive Behavioural Therapy Skills Questionnaire (CBTSQ)
  Intervention participants only. The CBTSQ is a 16-item maternal-report measure designed to assess cognitive and behavioural skills acquisition. Each item is scored on a 5-point scale, and total scores range from 16-80. Higher cognitive restructuring and behavioural activation scores predict reduction of overall psychiatric symptoms and depression.
Major Life Stress in the Past 12 Months | Baseline (T1)
  The Antenatal (Psychosocial) Risk Questionnaire (ANRQ) will be used to measure this outcome. The ANRQ is a 12-item self-report measure of psychosocial risk factors associated with increased risk for perinatal depression. One of the risk factors measured in the ANRQ is major life stress in the past 12 months, which would be considered job loss, separation, or bereavement. The ANRQ will also be used to assess additional risk factors for developing postpartum depression, including single marital status, a history of physical or sexual abuse, and/or poor social support. Scores on the ANRQ range from 5 to 60, with scores over 23 or higher used to identify women at increased risk for development of depression.
Socioeconomic Disadvantage | Baseline (T1)
  The Canadian Household Low Income Cut-Off (LICOs) Before Tax score will be calculated to determine socioeconomic status. The LICOs are income thresholds below which a family will likely devote a larger share of its income on the necessities of food, shelter and clothing than the average family. These thresholds are estimated by Statistics Canada to help identify Canadians who are likely to be substantially worse off than the average. LICOs vary by 7 family sizes and 5 different populations in terms of the area of residence.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Van Lieshout, MD, PhD, Principal Investigator — McMaster University
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Boland Z, Lloyd N, Drage J, Serrano-Lomelin J, Bieling P, Streiner D, Van Lieshout RJ. One-Day Online Cognitive Behavioral Therapy-Based Workshops for the Prevention of Postpartum Depression: A Randomized Controlled Trial. J Clin Psychiatry. 2025 Apr 16;86(2):24m15674. doi: 10.4088/JCP.24m15674. PMID 40257965